CLINICAL TRIAL: NCT07084051
Title: Intervention to Improve Medication Adherence Among Stroke Survivors in Rural Kentucky
Brief Title: Improve Medication Adherence Among Stroke Survivors in Rural Kentucky
Acronym: I-MAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hend Mansoor (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Hend Mansoor, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101375; 1P50MD019476-01 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stroke (CVA) or Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke Survivors (Experimental): self-management program with an an educational session and an individually-tailored session on medication adherence.
  Interventions: Behavioral: I-MAS

INTERVENTIONS:
Behavioral: I-MAS — Participants will receive a one-to one session with the pharmacy technician that involves two parts; the first part include education on ischemic stroke and risk factors such as practical strategies to improve hypertension control (i.e., appropriately taking medications, necessity of treatment, and consequences of not taking medicine, etc., making healthier dietary choices, exercising regularly, smoking cessation, alcohol intake, and managing blood sugar. The second part involves an interview to collect information on socio-demographics, clinical factors, co-morbidities, medications, and medication adherence barriers. During the second part of the session, the pharmacy technician will identify barriers to medication adherence for secondary prevention of stroke medications including antihypertensives, antithrombotic agents, and statins. The pharmacist will collaborate with the pharmacy technician to develop an action plan to address medication adherence barriers
  Other Names: Improve Medication Adherence Among Stroke Survivors

SUMMARY:
To test the feasibility and promise of a combined intervention provided by community health worker (CHW) in collaboration with pharmacy technician and pharmacist to improve hypertension and long-term stroke outcomes by identifying and reducing barriers to medication adherence among ischemic stroke survivors. This collaborative intervention involves a self-management program including an educational session on practical strategies to improve hypertension control (i.e., appropriately taking medications, necessity of treatment, and consequences of not taking medicine, etc.), complemented by individually-tailored sessions to identify and address barriers to medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with history of ischemic stroke or transient ischemic attack (TIA) in the past 2 years
* residing in a rural county in Kentucky

Exclusion Criteria:

* significant aphasia
* cognitive impairment
* a terminal illness
* other neurologic deficits that would impede from providing informed consent or meaningfully participate in the one-to-one sessions.
* a prior aneurysmal subarachnoid hemorrhage and or aneurysm, cerebral venous sinus thrombosis, vasculitis, blood clotting disorder due to genetic causes
* if the patient does not take any secondary preventative medications

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Medication Adherence Questionnaire | Baseline and at 3 months
  Medication adherence is measured using a 12-item questionnaire that determines how often medications are missed. Scores range from 12 to 48 with lower scores indicating better adherence

CONTACTS AND LOCATIONS:
Overall Officials: Hend Mansoor, PharmD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT07084051/ICF_000.pdf